CLINICAL TRIAL: NCT05492864
Title: Correction of Anterior Open Bite With Skeletally Anchored Extrusion Arch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9148620
Record Dates: First submitted 2022-07-24; First posted 2022-08-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-07

CONDITIONS: Anterior Openbite Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open bite with extrusion arch (Experimental): single arm study, measures will be recorded before and after
  Interventions: Procedure: extrusion of the anterior teeth

INTERVENTIONS:
Procedure: extrusion of the anterior teeth — sectional leveling and alignment of the teeth, then using of the extrusion arch as an overlay wire to treat the open bite

SUMMARY:
This study will aim to evaluate the effect of skeletally anchored extrusion arch on the dentofacial structures in patients with anterior open bite (AOB).

DETAILED DESCRIPTION:
This study will be a prospective clinical study. All the patients will be treated with 0.022 inch slot Roth metal brackets. Orthodontic bands will be cemented to the maxillary first molars. Both maxillary and mandibular teeth, will be sectionally leveled and aligned with superelastic Ni-Ti archwires.

A buccal stiff sectional wire from the first molar to the canine will be added for anchorage reinforcement. Extrusion will be done by inverting a 0.017 × 0.025-inch Connecticut intrusion archwire and inserting it in the molar auxiliary tubes upside-down and miniscrew will be tied to the molar bands to act as additional indirect anchorage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a class I or a mild class II dental relationship.
2. All permanent teeth are erupted except the third molars.
3. Mild to moderate open bite is present.
4. Normal or minimally increased facial height.
5. Low lip line.
6. No or Mild crowding.

Exclusion Criteria:

1. Patients with skeletal open bite.
2. Posterior cross bite.
3. Trauma to the maxillary incisor.
4. Patients in need to extraction due to sever crowding.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Mean change in the overbite and overjet "Amount of open bite closure". -Measurements will be done on pretreatment and posttreatment digital study models in millimeters(mm) | one year
  Amount of open bite closure measurement will help to know the effect of skeletally anchored extrusion arch on the treatment of anterior open bite
  * Mean change will be measured on pretreatment and posttreatment digital study models by measuring the vertical linear distance between the mesiodistal midpoint of the incisal edge of the uppermost vertically erupted upper central incisors and a horizontal plane projected on the lower central incisor(overbite) in millimeters(mm).
  * Also mean change will be measured on pretreatment and posttreatment digital study models by measuring the horizontal linear distance between the incisal edge of the most protruded upper central incisor and a frontal plane projected on the lower central incisor (overjet) in millimeters (mm).

SECONDARY OUTCOMES:
Mean change in the Antero-posterior position of permanent maxillary first molar. -Measurements will be done on pretreatment and posttreatment digital study models in millimeters(mm) | one year
  * Mean change in the Antero-posterior position of permanent maxillary first molar will help to know the effect of skeletally anchored extrusion arch on the posterior teeth.
  * Change will be measured on pretreatment and posttreatment digital study models by measuring the linear distance between the mesial surface of the upper first molar and a line joining the medial end of the two third rugae, the mean between the right and left sides will be used in millimeters(mm)
  * Also will be measured on pretreatment and posttreatment digital study models by measuring the horizontal linear distance between the mesiobuccal cusp of upper first molar and mesiobuccal groove of lower first molar, the mean between the right and left sides will be used in millimeters (mm).
Changes that occur in the dentoalveolar vertical development of the upper and lower anterior teeth. -Measurements will be done on pretreatment and posttreatment digital study models in millimeters(mm) | one year
  * Changes that occur in the dentoalveolar vertical development of the upper and lower anterior teeth will help to know the effect of skeletally anchored extrusion arch on the vertical development of the anterior teeth.
  * Change will be measured on pretreatment and posttreatment digital study models by measuring The perpendicular vertical distance from a point between the central incisors at the level of the alveolar process to the occlusal plane from the frontal view, the occlusal plane was determined by three points: mesiobuccal cusp tip of the right and left first permanent molars and cusp tip of the right first premolar in millimeters (mm).
  * Also will be measured on pretreatment and posttreatment digital study models by measuring the vertical distance between the incisal edge and gingival margin of the central incisor along its labial surface, the mean between the right and left sides will be used in millimeters(mm).
Changes that will occur in the upper and lower arch length, perimeter and intermolar width. -Measurements will be done on pretreatment and posttreatment digital study models in millimeters(mm) | one year
  * This outcome will help to know the effect of skeletally anchored extrusion arch on the upper and lower arch length, perimeter and intermolar width.
  * Change will be measured on pretreatment and posttreatment digital study models by measuring the perpendicular distance between a line connecting the mesial aspects of the permanent first molars and the contact point between the central incisors (arch length) in millimeters(mm), measuring the sum of four segments: from the mesial surface of the permanent first molar to the mesial contact point of the canine and then to the contact point of the central incisors, measured on the right and left sides (arch perimeter)in millimeters (mm) and measuring the linear distance between right and left first permanent molar (intermolar width) in millimeters (mm).
Skeletal, dental and soft tissues changes . Measurements will be done on pretreatment and posttreatment lateral cephalometric radiographs in degree (°) | one year
  * This outcome will help to know the effect of skeletally anchored extrusion arch on the dentofacial structures in patients with anterior open bite.
  * Measurements will be done on pretreatment and posttreatment lateral cephalometric radiographs:
  * SNA(°)/SNB(°)/ANB(°) will show changes in skeletal antero-posterior relationship between maxilla and mandible.
  * MP(Me-GO)-SN(°)/Palato-mandibular plane(°)/FH-OP(°)/FH-PP(°)/Gonial angle(°) will show skeletal vertical changes.
  * Occlusal plane- SN (°) will show dental vertical changes.
  * L1-MP(°)(IMPA)/U1-PP(°)/Interincisal angle(°) will show dental incisor inclination.
  * Nasolabial angle(°) will show Soft tissues changes.
Skeletal, dental and soft tissues changes . Measurements will be done on pretreatment and posttreatment lateral cephalometric radiographs in millimeters (mm) | one year
  * This outcome will help to know the effect of skeletally anchored extrusion arch on the dentofacial structures in patients with anterior open bite.
  * Measurements will be done on pretreatment and posttreatment lateral cephalometric radiographs:
  * Witts(mm) will show changes in skeletal antero-posterior relationship between maxilla and mandible.
  * ALFH(ANS-Me)(mm)/A-ANS(mm)/N-Me(mm)/Co-GO(mm) will show skeletal vertical changes.
  * U6-PP(mm)/U1-pp(mm)/L6-MP(mm)/L1-MP(mm) will show dental vertical changes.
  * U1-Eplane(mm)/L1-Eplane(mm) will show Soft tissues changes.
Change in the smile of the patients through measuring mean change in the lenght of the upper lip, amount of incisors and gum exposure. Measurements will be done on pretreatment and posttreatment photographs in millimeters (mm). | one year
  This outcome will help to know the effect of extrusion of the anterior teeth on the smile of the patients.
  Pretreatment and posttreatment extraoral photographs will be taken, including a close-up photograph with a ruler while the patient is smiling.
Stability of the treatment after 1, 2 and 3year(s) through measuring mean change in the overbite. Measurements will be done on digital study models in millimeters(mm) | Two year, three and four year.
  This outcome will help to know the stability of the technique of using of skeletally anchored extrusion arch in the treatment of anterior open bite patients.
  -stability will be measured on posttreatment after 1, 2 and 3 years posttreatment digital study models by measuring the vertical linear distance between the mesiodistal midpoint of the incisal edge of the uppermost vertically erupted upper central incisors and a horizontal plane projected on the lower central incisor(overbite) in millimeters(mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No